CLINICAL TRIAL: NCT05133973
Title: Effectiveness and Safety Study to Investigate the Improved FiberSense Continuous Glucose Monitoring System in Diabetic Patients
Brief Title: Feasibility Study of a Transdermal Continuous Glucose Monitoring (CGM) System in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeSense GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: P-4.7-C-01
Record Dates: First submitted 2021-11-05; First posted 2021-11-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2022-10

CONDITIONS: Diabetes
Keywords: diabetes management; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Subjects will wear 3 FiberSense systems (2x arm and 1x abdomen) and one comparator. The subjects will participate in six clinic in-house sessions on Day 00, 3x between days 01-07, on Days 21 and 28. There will be safety visit at Day 14.
  Finger pricking at home use will be intensified during days 00-07.
  Interventions: Device: FiberSense CGM
- Cohort B (Experimental): Subjects will wear 3 FiberSense systems (2x arm and 1x abdomen) and one comparator. The subjects will participate in six clinic in-house sessions on Day 00, 4x between days 07-14 and on Day 28. There will be safety visit at Day 21.
  Finger pricking at home use will be intensified during days 07-14.
  Interventions: Device: FiberSense CGM

INTERVENTIONS:
Device: FiberSense CGM — FiberSense system, a novel CGM system, based on a fiber-optical sensor placed through the dermis of the patient.

SUMMARY:
A single centered, prospective, double blinded study enrolling 12 Type I diabetic patients (+ up to 4 replacements) in two cohorts. Patients will wear multiple FiberSense CGM systems for 28 days, with total duration of the participation up to 8 weeks (screening + active phase + follow up).

The primary aims of the study are assessment of the safety and tolerability of the FiberSense CGM system during the wearing time together with characterization of the system performance when compared to capillary blood samples.

DETAILED DESCRIPTION:
The FiberSense system is intended to be used by diabetic patients in a home use setting as a CGM system using the interstitial fluid (ISF) glucose as an indicator of blood glucose levels.The purpose of this study is to assess the performance of FiberSense system across the glucose measurement ranges as compared with a laboratory standard reference method in diabetic patients (Type I) during in-clinic glucose challenge sessions. At the same time and also at home use the blood glucose values are recorded by comparator system and self-monitoring blood glucose system (SMBG). The safety aspects are also investigated during the wearing time of 28 days.

The two cohorts differ in the measurement scheduled, with intensive measurement week either at week 1 (cohort A) or week 2 (cohort B).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 and < 65 years old.
2. Diabetes mellitus type I requiring insulin in the management of glucose control for at least one year prior to enrollment.
3. Women who are not pregnant, lactating or planning a pregnancy during their participation in the clinical study. If of child bearing potential, the patient must agree to abstain from sexual intercourse or use reliable forms of contraception (e.g. condom or diaphragm with spermicide or oral contraceptives) to prevent pregnancy for the length of the clinical study.
4. Willingness, ability and commitment to comply with the testing, procedure and follow-up outlined in this protocol including (but not limited to) frequency of clinic visits, use of pre-specified glucose monitoring devices.
5. In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a good study candidate.
6. For the time of the wearing phase willingness to abstain from taking a sauna, bathing, swimming, diving and contact sport activities.
7. Fully vaccinated with EMA approved vaccine against SARS-COV-2 virus or recovered from Covid-19 disease, (status vaccinated or recovered according to current Corona regulations as recommended by STIKO). If applicable, a negative result of a current Corona test (depending on the guidelines of the study center).
8. Written informed consent to participate in the study provided by the patient.

Exclusion Criteria:

1. Persons who use medication containing icodextrine or maltose and which can result in icodextrine or maltose present in blood (dialysis solutions, antibody medications etc.), anamnesis based.
2. Persons on peritoneal dialysis.
3. History of significant hypoglycemia unawareness, or a history of severe hypoglycemia (requiring emergency medical intervention) within the last 6 months.
4. Currently pregnant, as demonstrated by a positive pregnancy test at screening and/or Day00 prior to enrolment.
5. Any active acute or chronic infectious disease that, in the opinion of the investigator, might interfere with the performance of this study or would pose an excessive risk to study staff (e.g., Hepatitis B and C, HIV, Covid-19).
6. Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
7. Have a known allergy to medical-grade adhesives, or known hypersensitivity to any of the products used in the study.
8. Blood donation of more than 500 ml within the last three months or hematocrit value <30% or > 50%.
9. Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
10. Has a MRI scan, CT scan, diathermy or a flight scheduled during the proposed study participation.
11. Has vaccination/booster against COVID-19 scheduled during or less than 2 weeks prior to the proposed study participation.
12. An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Performance of the FiberSense system as compared with laboratory gold standard reference (LGSR) | 6 measurements within 28 days
  Point accuracy of the FiberSense system as determined by proportion of CGM readings within ≤15% of the LGSR reading for blood glucose levels >100 mg/dl, and within ≤15 mg/dl of the LGSR reading for blood glucose levels ≤100 mg/dl (15/15%), for paired samples taken during the in-clinic sessions.
Incidence and severity of device related adverse events (ADE) | 28 days
  Incidence of reported ADE with focus on number of patients experiencing serious ADE, evaluated according Draize's scale (0 to 4 - for none to severe findings)

SECONDARY OUTCOMES:
FiberSense System agreement to LGSR within different glucose ranges | 6 measurements within 28 days
  The percentage of FiberSense CGM system readings within metrics 20/20%, 30/30%, 40/40% and greater than 40% of the laboratory reference values
Point Clinical accuracy (Consensus and Surveillance Error Grid) | 6 measurements within 28 days
  Analyze the proportion of readings in each region of two Grids. Readings in various regions are considered from clinically accurate or with clinically acceptable accuracy to inaccurate to various degrees.
Accuracy of glucose rate of change of FiberSense System during glucose excursions | 6 measurements within 28 days
  Mean and Median Absolute Relative Differences (MARD, MedRD) of FiberSense measured glucose from laboratory reference values, evaluated at various glucose dynamics
Agreement and accuracy relative to SMBG readings at home use | 6 measurements within 28 days
  Performance of FiberSense System evaluated as percentage of system readings within 15%, 20%, 30% and 40% of SMBG values
Precision of the FiberSense System (PARD) for arm-arm and arm-abdomen positions | 6 measurements within 28 days
  Precision Absolute Relative Difference (PARD) of two simultaneously worn FiberSense Systems by one patient, for same body parts and two different insertion sites
FiberSense System stability | weekly during 28 days
  Percentage of FiberSense System readings within various % of the LGSR values
FiberSense System Longevity | 28 days
  Duration of use of the individual FiberSense devices
User satisfaction questionnaire score | after 28 days
  Subjective impression of the patients assessed by 5-point Likert scale (1 - strongly agree to 5 - strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Freckmann, Dr.med., Principal Investigator — Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm
Locations (1):
- Institut für Diabetes-Technologie, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No